CLINICAL TRIAL: NCT02244333
Title: ALNA® - AWB in Pre-treated Patients With BPS
Brief Title: Efficacy, Tolerability and Safety of ALNA® in Patients With Benign Prostatic Syndrome (BPS)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 527.56
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with symptomatic BPS
  Interventions: Drug: ALNA®

INTERVENTIONS:
Drug: ALNA®

SUMMARY:
Study to assess efficacy, tolerability and safety parameters of a one month ALNA® - treatment after switch from Terazosin-treatment

ELIGIBILITY:
Inclusion Criteria:

* Suffering from BPS symptoms
* Preceding treating with Terazosin for at least one month
* IPSS sum score >= 8 points prior to treatment start with ALNA® or complaints due to BP reduction by Terazosin
* Indication for a switch to treatment with ALNA® according to its Summary of Product Characteristics (SPC) for a minimum period of one month

Exclusion Criteria:

* Patients fulfilling one of the general or specific contraindications listed in the ALNA® SPC, particularly patients with known hypersensitivities against tamsulosin hydrochloride or any other ingredients of the product, orthostatic dysregulation or severe liver insufficiency could not be included in the Post Marketing Surveillance (PMS) study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic BPS, who switched for ALNA® after preceding Terazosin therapy recruited at urologists
Sampling Method: Non-Probability Sample
Enrollment: 4575 (Actual)
Dates: Start 2004-02; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in International Prostatic Symptom Score (IPSS) by means on patient questionnaire | Baseline, after 1 month
Change of Quality of Life (QoL) Index by means on patient questionnaire | Baseline, after 1 month
Global comparative assessment of Terazosin and ALNA® treatment by investigator on a 3 point-scale | after 1 month

SECONDARY OUTCOMES:
Change from Baseline in maximum urinary flow rate (Qmax) | Baseline, after 1 month
Change from Baseline in residual urinary volume | Baseline, after 1 month
Change from Baseline in blood pressure | Baseline, after 1 month
Change from Baseline in Pulse rate (bpm) | Baseline, after 1 month
Change in complications due to low blood pressure | Baseline, after 1 month
  Patient is asked for complications (weakness, dizziness, nausea)
Global assessment of efficacy by investigator on 4-point scale | after 1 month
Global assessment of tolerability by investigator on 4-point scale | after 1 month
Global assessment with BPS- treatment by investigator on a 4-point scale | Baseline, after 1 month
  Switch from Terazosin therapy to ALNA®